CLINICAL TRIAL: NCT06597669
Title: Comparison of the Treatment Outcomes of the Conventional Stainless Steel Crown Restorations and the Hall Technique in the Treatment of Carious Primary Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hue University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Le Van Nhat Thang, Lecturer, Hue University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H2024/097
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Caries,Dental
Keywords: Dental caries; Primary molars; Stainless steel crowns
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Technique (Experimental): A stainless steel crown will place on a carious primary molar after preparation
  Interventions: Procedure: Placement of stainless steel crowns on primary molars
- Hall technique (Experimental): A stainless steel crown will place on a carious primary molar without local anesthesia caries removal or any preparation
  Interventions: Procedure: Placement of stainless steel crowns on primary molars

INTERVENTIONS:
Procedure: Placement of stainless steel crowns on primary molars — Preformed metal crowns have been placed to treat caries in primary molars

SUMMARY:
Stainless steel crowns have shown high success in restoring carious primary molars over a longer period of time than conventional restorations. This study aims to evaluate the treatment effectiveness of conventional SSCs restoration and Hall technique in treating carious primary molars

ELIGIBILITY:
Inclusion Criteria:

1. Agree and voluntarily participate in the research (with the patient's parent/guardian consent for participation)
2. Children have a primary molar with at least 2 carious lesions corresponding to International Caries Detection and Assessment System (ICDAS) scores 4 or at least 1 carious lesion corresponding to ICDAS scores 5 and 6.

Exclusion Criteria:

1. Children with systemic diseases such as immunodeficiency, cardiovascular disease, or bleeding disorders.
2. Children are allergic to nickel and resin.
3. Children unable to return for recall visits.
4. Primary molar has signs of pulpal/periapical diseases (irreversible pulpitis, pulp necrosis, loosening, fistula, or abscess).
5. Children are undergoing orthodontic treatment with fixed or removable appliances.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Failure of stainless steel crowns | 3 months
  Level 1 failures was considered when there were any signs of failure related to SSCs. Level 2 failures was considered when there were any signs of related pulpal and periapical pathology. Success was considered when Level 1 and 2 failures were absent.
Failure of stainless steel crowns | 6 months
  Level 1 failures was considered when there were any signs of failure related to SSCs. Level 2 failures was considered when there were any signs of related pulpal and periapical pathology. Success was considered when Level 1 and 2 failures were absent.
Failure of stainless steel crowns | 9 months
  Level 1 failures was considered when there were any signs of failure related to SSCs. Level 2 failures was considered when there were any signs of related pulpal and periapical pathology. Success was considered when Level 1 and 2 failures were absent.
Failure of stainless steel crowns | 12 months
  Level 1 failures was considered when there were any signs of failure related to SSCs. Level 2 failures was considered when there were any signs of related pulpal and periapical pathology. Success was considered when Level 1 and 2 failures were absent.

SECONDARY OUTCOMES:
Occlusal contact | 0 months
  Occlusal contact was assessed as follows: normal occlusion or rised occlusion.
Occlusal contact | 3 months
  Occlusal contact was assessed as follows: normal occlusion or rised occlusion.
Occlusal contact | 6 months
  Occlusal contact was assessed as follows: normal occlusion or rised occlusion.
Occlusal contact | 9 months
  Occlusal contact was assessed as follows: normal occlusion or rised occlusion.
Occlusal contact | 12 months
  Occlusal contact was assessed as follows: normal occlusion or rised occlusion.
Periodontal health | 0 months
  * Plaque index 0 = No plaque in the gingival area.
    1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
    2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
    3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
  * Gingival index 0 = Normal gingiva
    1. = Mild inflammation - slight change in color, slight oedema. No bleeding on probing
    2. = Moderate inflammation-redness, oedema and glazing. Bleeding on probing
    3. = Severe inflammation - marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.
Periodontal health | 3 months
  * Plaque index 0 = No plaque in the gingival area.
    1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
    2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
    3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
  * Gingival index 0 = Normal gingiva
    1. = Mild inflammation - slight change in color, slight oedema. No bleeding on probing
    2. = Moderate inflammation-redness, oedema and glazing. Bleeding on probing
    3. = Severe inflammation - marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.
Periodontal health | 6 months
  * Plaque index 0 = No plaque in the gingival area.
    1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
    2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
    3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
  * Gingival index 0 = Normal gingiva
    1. = Mild inflammation - slight change in color, slight oedema. No bleeding on probing
    2. = Moderate inflammation-redness, oedema and glazing. Bleeding on probing
    3. = Severe inflammation - marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.
Periodontal health | 9 months
  * Plaque index 0 = No plaque in the gingival area.
    1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
    2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
    3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
  * Gingival index 0 = Normal gingiva
    1. = Mild inflammation - slight change in color, slight oedema. No bleeding on probing
    2. = Moderate inflammation-redness, oedema and glazing. Bleeding on probing
    3. = Severe inflammation - marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.
Periodontal health | 12 months
  * Plaque index 0 = No plaque in the gingival area.
    1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
    2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
    3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
  * Gingival index 0 = Normal gingiva
    1. = Mild inflammation - slight change in color, slight oedema. No bleeding on probing
    2. = Moderate inflammation-redness, oedema and glazing. Bleeding on probing
    3. = Severe inflammation - marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Hue University of Medicine and Pharmacy, Huế, Thừa Thiên Huế Province, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Will plan to share information when finishing study
Supporting Information: Study Protocol, SAP, CSR